CLINICAL TRIAL: NCT02816983
Title: A Phase II Evaluation of SBRT in Oligometastatic Castration-Refractory Prostate Cancer and Immunogenicity of SBRT
Brief Title: SBRT for Oligometastatic Castration-Refractory Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sean S. Park, PI, Mayo Clinic
Other Study IDs: 16-000785; CA200551 (Other: NIH/NCI)
Record Dates: First submitted 2016-06-25; First posted 2016-06-29 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SBRT for oligometastatic prostate cancer
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT
  Other Names: Stereotactic ablative radiotherapy (SABR)

SUMMARY:
Castration-resistant prostate cancer patients with rising prostatic specific antigen (PSA) are eligible for this study. 11C-Choline PET/CT will be used to identify metastatic lesions. Patients with <=3 metastatic lesions will receive stereotactic body radiotherapy (SBRT) as definitive treatment. Blood draws will be taken to monitor the development of anti-prostate cancer immunity

ELIGIBILITY:
Inclusion Criteria:

* Patients must be receiving standard of care SBRT as outlined in the Universal Content Management (UCM) Procedure Manual (http://mayocontent.mayo.edu/radoncology/categories/index.html)
* Age ≥ 18 years.
* Metastatic castration-refractory prostate cancer patients with ≤ 3 lesions identified on standard imaging and/or choline PET/CT within 60 days of registration
* Castrate levels of testosterone
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2 (Appendix I).
* Life expectancy > 6 months

Exclusion Criteria:

Emergent cord compression for spinal metastases

* Severe, active co-morbidity, defined as follows:

  1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration
  2. Transmural myocardial infarction within the last 6 months prior to registration
  3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  4. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration
  5. Severe hepatic disease, defined as a diagnosis of Child-Pugh Class B or C hepatic disease.
  6. HIV positive with Cluster Differentiation 4 (CD4) count < 200 cells/microliter. Note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count ≥ 200 cells/microliter within 30 days prior to registration. Note also that HIV testing is not required for eligibility for this protocol.
  7. End-stage renal disease (i.e., on dialysis or dialysis has been recommended).
* Metastases located within 3 cm of the previously irradiated structures:

  1. Spinal cord previously irradiated to > 40 Gy
  2. Brachial plexus previously irradiated to > 50 Gy
  3. Small intestine, large intestine, or stomach previously irradiated to > 45 Gy
  4. Brainstem previously irradiated to > 50 Gy
  5. Lung previously irradiated with prior V20Gy > 30%

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be receiving standard of care SBRT
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
PSA-progression free survival | 1 year
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sean S Park, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhang H, Orme JJ, Abraha F, Stish BJ, Lowe VJ, Lucien F, Tryggestad EJ, Bold MS, Pagliaro LC, Choo CR, Brinkmann DH, Iott MJ, Davis BJ, Quevedo JF, Harmsen WS, Costello BA, Johnson GB, Nathan MA, Olivier KR, Pisansky TM, Kwon ED, Dong H, Park SS. Phase II Evaluation of Stereotactic Ablative Radiotherapy (SABR) and Immunity in 11C-Choline-PET/CT-Identified Oligometastatic Castration-Resistant Prostate Cancer. Clin Cancer Res. 2021 Dec 1;27(23):6376-6383. doi: 10.1158/1078-0432.CCR-21-2510. Epub 2021 Sep 30. PMID 34593526
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials